CLINICAL TRIAL: NCT07400588
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Study of the Safety and Tolerability of Aleniglipron in Adult Participants With Type 2 Diabetes Mellitus Living With Obesity or Overweight
Brief Title: Aleniglipron Phase 2 in Type 2 Diabetes Mellitus
Acronym: GSBR-1290
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gasherbrum Bio, Inc., a wholly owned subsidiary of Structure Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GSBR-1290-17
Record Dates: First submitted 2025-10-28; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Obese; Obesity; Obesity Type 2 Diabetes Mellitus; Weight Loss
Keywords: Obese; obesity; Obesity Type 2 Diabetes; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Participants will receive aleniglipron administered orally (Experimental): Drug aleniglipron administered orally
  Interventions: Drug: Aleniglipron
- Arm 2: Participants will receive a placebo administered orally (Experimental): Drug placebo administered orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aleniglipron — Drug aleniglipron administered orally
  Arms: Arm 1: Participants will receive aleniglipron administered orally
Drug: Placebo — Drug placebo administered orally
  Arms: Arm 2: Participants will receive a placebo administered orally

SUMMARY:
The purpose of this study is to assess the safety and tolerability of aleniglipron at doses up to 240 mg once daily (QD) in participants with T2DM who are living with obesity (body mass index [BMI] ≥ 30 kg/m2) or overweight (BMI ≥ 27 kg/m2).

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* A diagnosis of T2DM of ≥6 months,
* Hemoglobin A1c (HbA1c) ≥6.5% to ≤10% at Screening
* Have a BMI ≥27.0 kg/m2

Exclusion Criteria:

* Are currently receiving or planning to receive treatment for diabetic retinopathy and/or macular edema. All participants must have a photo fundoscopy, optical coherence tomography, or slit lamp assessment prior to randomization and within the last 12 months to confirm the absence or stable status of diabetic retinopathy and/or macular edema.
* Present or planned use of any drug that could interfere with glucose levels
* Self-reported change in body weight >5 kg (11 pounds) within 3 months before screening
* Have prior or planned surgical treatment for obesity (excluding liposuction or abdominoplasty, if performed >1 year prior to Screening)
* Have or plan to have endoscopic and/or device-based therapy for obesity or have had device removal within the last 6 months prior to Screening, including, but not limited to, mucosal ablation, gastric artery embolization, intragastric balloon, and duodenal-jejunal endoluminal liner

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity and relationship of AEs/SAEs | Baseline to week 38
Assessment of vital signs | Baseline to week 38
  Number of Participants with Clinically Significant Change from Baseline in Vital Signs: including Systolic and Diastolic Blood Pressure, Heart Rate, and temperature.
Assessment of laboratory measures | Baseline to week 38
  Number of Participants with Clinically Significant Change from Baseline in Laboratory Parameters: including hematology, serum chemistry, coagulation
Assessment of Electrocardiograms (ECG) | Baseline to week 38
  Number of Participants with Clinically Significant Change from Baseline in Electrocardiogram (ECG) Parameters: Common ECG-related variables will be assessed, including but not limited to: ventricular heart rate, PR interval, QRS duration, QT interval, and QTcF

SECONDARY OUTCOMES:
Absolute change in body weight from Baseline | Baseline to week 39
Percent change in body weight from Baseline | Baseline to week 39
Change in HbA1c from Baseline | Baseline to week 39
Change in fasting plasma glucose from Baseline | Baseline to week 39
PK parameters including but not limited to AUC | Baseline to week 39
PK parameters including but not limited to Cmax | Baseline to week 39
TPK parameters including but not limited to Tmax | Baseline to week 39
PK parameters including but not limited to Ctrough | Baseline to week 39

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Research Site, Anniston, Alabama
  - Research Site, Lake Forest, California
  - Research Site, Lomita, California
  - Research Site, Hazelwood, Missouri
  - Research Site, Columbus, Ohio
  - Research Site, Moncks Corner, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, DeSoto, Texas
  - Research Site, Houston, Texas
  - Research Site, Mesquite, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Tomball, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address a specific research question in an approved data sharing request
Supporting Information: Study Protocol
Time Frame: Data sharing requests will be considered beginning 36 months after the study publication (manuscript accepted for publication) and either 1) the product has been granted marketing authorization in at least two regulatory jurisdictions, or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Researchers will submit a request containing the research objectives, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). Gasherbrum Bio, Inc. does not grant external requests for individual de-identified patient data for the following purposes:
  * Re-evaluating safety and efficacy end points already addressed in the product labelling,
  * Assessing safety or efficacy for an indication in current development Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a panel of external advisors. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement.